CLINICAL TRIAL: NCT04256850
Title: Teaching Novel Values-Based Skills to Improve Long-Term Weight Loss: A Randomized Trial Examining the Efficacy of a Weight Loss Maintenance Intervention Based on Acceptance and Commitment Therapy
Brief Title: Teaching Novel Values-Based Skills to Improve Long-Term Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK120731 (NIH)
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Acceptance and Commitment Therapy; Professional Autonomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (ACT) (Experimental): Focuses on addressing cognitive and emotional barriers to successful weight loss maintenance.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Self-Regulation (SR) (Experimental): Focuses on using self-monitoring and self-reinforcement techniques to improve weight loss maintenance.
  Interventions: Behavioral: Self-Regulation (SR)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Teaches acceptance, mindfulness, and values-based skills
  Arms: Acceptance and Commitment Therapy (ACT)
Behavioral: Self-Regulation (SR) — Teaches monitoring and reinforcement strategies designed to improve motivation and adherence to positive weight loss behavioral prescriptions.
  Arms: Self-Regulation (SR)

SUMMARY:
This NIDDK funded R01 project is a randomized controlled clinical trial to compare the efficacy of an intervention based on Acceptance and Commitment Therapy (ACT) and a Self-Regulation (SR) intervention on weight loss maintenance over a 30-month period. All participants will first complete a well-validated online weight loss intervention (months 1-3 of the study). Participants who lose ≥4 kilograms of initial weight will then be randomly assigned to receive ACT or SR, with both conditions consisting of face-to-face, group-based intervention meetings and weekly email contact for 6 months.

DETAILED DESCRIPTION:
Obesity is a major public health problem, and although short-term weight loss is achievable, individuals often regain the majority of weight that was lost. Current approaches have adjusted behavioral prescriptions and lengthened treatment contact in an effort to address this problem, with modest effect. This NIDDK funded R01 project is a randomized controlled clinical trial to compare the efficacy of an intervention based on Acceptance and Commitment Therapy (ACT) and a Self-Regulation (SR) intervention on weight loss maintenance over a 30-month period. All participants will first complete a well-validated online weight loss intervention (months 1-3 of the study). Participants who lose ≥4 kilograms of initial weight will then be randomly assigned to receive ACT or SR, with both conditions consisting of face-to-face, group-based intervention meetings and weekly email contact for 6 months. The ACT intervention will target a novel theoretically derived intervention target, values-consistent behavior, which will help align weight loss goals with personal values and foster internal motivation to continue with weight control efforts. Assessments will be at baseline, post-weight loss/pre-randomization, and then 6, 12, 18, 24, and 30-month follow-up (months from randomization). This project will be conducted at the Weight Control and Diabetes Research Center (WCDRC). The WCDRC is part of the Centers for Behavioral and Preventive Medicine at The Miriam Hospital in Providence, Rhode Island, and the Department of Psychiatry and Human Behavior at the Alpert Medical School of Brown University. This study is significant because it addresses weight loss maintenance - a critical barrier to treating obesity - and results of the study could be used to improve long-term weight loss outcomes and associated health benefits for treatment seeing overweight and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* English language fluent and literate at the 6th grade level
* Body mass index (BMI) between 27.5 and 45 kg/m-squared
* Able to walk 2 city blocks without stopping
* Has reliable access to a computer with internet access

Exclusion Criteria:

* Currently participating in another weight loss program
* Currently taking weight loss medication
* Has lost ≥5% of body weight in the 6 months prior to enrolling
* Has been pregnant within the 6 months prior to enrolling
* Plans to become pregnant within 18 months of enrolling
* Has a heart condition, chest pain during periods of activity or rest, or loss of consciousness in the 12 months prior to enrolling
* Has any medical condition that would affect the safety of participating in unsupervised physical activity
* Has any condition that would result in inability to follow the study protocol, including terminal illness and untreated major psychiatric illness

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Weight Loss Maintenance | 30 months
  weight change from randomization to study end

SECONDARY OUTCOMES:
Waist Circumference | 30 months
  change in waist circumference from randomization to study end
Objectively Measured Physical Activity Minutes Per Week | 30 months
  change in objectively measured physical activity from randomization to study end as measured by 7 days of wearing Actigraph accelerometer device

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lillis, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data includes objective measurement of weight and height, physical activity, dietary intake, and self-report questionnaire data assessing values-consistent behavior, motivation, and use of weight control strategies. The final dataset will include self-reported demographic data. Research data from participants may be shared with the broader scientific community after publication. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that protecting the identities of participants is best achieved by enacting additional safeguards. We will therefore make data and documentation available only under a data-sharing agreement that provides for (1) a commitment to use the data for research purposes only; (2) a commitment to securing the data using appropriate computer technology; (3) a commitment to destroying or returning the data after analyses are completed; and (4) a commitment not to attempt to identify participants individually.
Time Frame: After data analysis for the study is complete.

REFERENCES:
- [Derived] Emerson JA, Schumacher LM, Bond DS, Thomas JG, Lillis J. Physical activity changes during an automated online weight loss program. J Behav Med. 2023 Aug;46(4):680-688. doi: 10.1007/s10865-022-00383-6. Epub 2023 Jan 5. PMID 36602619